CLINICAL TRIAL: NCT01799213
Title: Discontinuing NSAIDs in Veterans With Knee Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IIR 11-113
Record Dates: First submitted 2013-02-22; First posted 2013-02-26 (Estimated); Results first posted 2019-12-16 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis; NSAID; Cognitive Behavioral Therapy
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Meloxicam; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active Treatment (Experimental): Eligible subjects will be randomized to Meloxicam 15 mg po per day (QD) vs placebo
  Interventions: Drug: Meloxicam 15 mg po QD
- Placebo (Placebo Comparator): Eligible subjects will be randomized to Meloxicam 15 mg po QD vs placebo
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Drug: Meloxicam 15 mg po QD — Eligible subjects will be take Meloxicam 15 mg po QD
  Arms: Active Treatment
Behavioral: Cognitive Behavioral Therapy — Subjects originally assigned to placebo will receive cognitive behavioral therapy for 10 weeks
  Arms: Placebo

SUMMARY:
Knee osteoarthritis (OA) is now recognized as a major health problem. It is the number one cause of lower extremity disability and has significant deleterious effects on quality of life. While there are numerous therapies available for knee OA, most have limited efficacy. Of particular concern, is the widespread use of nonsteroidal anti-inflammatory drugs (NSAIDs) for this disorder. Veterans, as a group, are at high risk for both gastrointestinal and cardiovascular NSAID-induced complications. In this study the investigators propose to examine whether replacing NSAIDs with cognitive behavioral therapy delivered by telephone is an effective strategy for Veterans with knee OA. Telephone-administered therapy is particularly appealing since Veterans with knee OA are more likely to have limited mobility. If successful, this program may result in significant cost-savings for both Veterans (decreased co-pays and transportation costs) and the VA (decreased hospitalizations due to NSAID induced toxicity).

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is a major cause of disability among Veterans and is the primary indication of knee replacement in the VA. Nonsteroidal anti-inflammatory drugs (NSAIDs) are the most commonly prescribed medications for knee OA. Though short-term studies have demonstrated that NSAIDs are more effective than placebo and acetaminophen, there are no long-term data supporting their use. This is of concern, because long-term use of NSAIDs is associated with significant morbidity and mortality. Guidelines have been published to improve safe use of NSAIDs; however, adherence to these evidence-based recommendations is low in the VA. There is therefore an important need to determine if the long-term use of NSAIDs offers any incremental benefit over safer alternatives. This is especially true for Veterans, a population at high risk for NSAID-induced toxicity.

Cognitive behavioral therapy (CBT) is an effective and safe treatment alternative for OA. This modality is becoming increasingly available in the VA for treatment of chronic pain as well as other chronic disorders such as depression, post-traumatic stress disorder and insomnia. CBT can be successfully administered over the telephone and thus stands to benefit Veterans living in more remote areas with limited access to hospital or community-based outpatient clinics.

In this study, the investigators propose to conduct a 2-phase randomized withdrawal trial (RWT). The trial will focus on recruiting Veterans with knee OA who have been using NSAIDs for at least 3 months.

In the first phase of the study, 544 Veterans with knee OA will be randomized to continue NSAIDs or to placebo for 4 weeks. This double-blind phase will enable us to infer whether placebo is non-inferior to continued NSAID use. In the second phase, subjects in the NSAIDs group will continue NSAIDs and those on placebo will stop taking the placebo and participate in a 10-week CBT program. The second, single-blind, phase will allow us to infer whether CBT is non-inferior to NSAIDs. All study data will be collected over the telephone thus enabling Veterans who have difficulty arranging transportation to the VA to participate.

The investigators will test for between-group differences in knee pain measured using the well-validated Western Ontario and McMaster Universities Osteoarthritis Index (primary outcome) at 4 and 14 weeks. The investigators will also test for between group differences in lower extremity disability, subjects' global impression of change and use of co-therapies (secondary outcomes). As recommended for non-inferiority trials, the investigators will perform both an intent to treat and per protocol analysis. Lastly, the investigators will estimate the potential cost-effectiveness of the CBT protocol compared with continued NSAID use.

Though it would be ideal for subjects randomized to the active study drug to continue their current NSAID, having the VA pharmacy formulate multiple different active drugs and maintaining the blind is not possible. Therefore, the investigators will include a 2-week run-in period where study subjects will replace their NSAID with meloxicam. Meloxicam was chosen as the study drug because it is the most commonly prescribed at the investigators' center and has a favorable safety profile compared to other NSAIDS.

If successful, the trial will improve the quality of care delivered to Veterans with chronic knee pain due to OA. The proposed strategy is particularly appealing because it replaces the widespread use of NSAIDs with a safer alternative, enables delivery of care to Veterans with limited access, and is likely to be cost saving.

ELIGIBILITY:
Inclusion Criteria:

Subjects will include those for whom a discontinuation trial of NSAIDs is most appropriate: 1) Veterans with knee pain despite NSAID use and/or 2) Veterans at relatively higher risk of NSAID toxicity 55-59 as ascertained by meeting 1 or more of the following 4 criteria:

* Answer affirmatively to the question: "Do you have some knee pain on most days over the past 3 months?"
* Have 1 or more risk factors for NSAID-induced nephrotoxicity (age greater than 60 years, atherosclerotic cardiovascular disease, current diuretic use, chronic renal insufficiency, congestive heart failure (New York Heart Association class I-II. Note, Class III and IV are excluded).
* Have 1 or more risk factors for NSAID-induced gastrointestinal toxicity (history of peptic ulcer disease, age > 65 years, concurrent use of daily ASA or corticosteroids), and are currently on a gastro-protective agent.
* Have 1 or more risk factors for NSAID-induced cardiovascular toxicity (prevalent cardiovascular disease, hypertension, hypercholesterolemia, diabetes, smoking, family history of early heart disease or age greater than 55 years for women).

In addition, subjects must:

* Be age 20 years or older. While the usual cut off for knee OA is approximately 40 years, the investigators chose to lower the age cutoff as younger Veterans have a higher than expected risk of OA (see B.1).
* Have radiographic evidence of knee OA reported in the VistA electronic system.
* Be using an NSAID (other than daily ASA) for knee pain on most days of the month for at least the past 3 months.
* Be able to understand and speak English and have a telephone.
* Be willing to engage in a CBT program, to discontinue (or replace) their NSAID, and to restrict co-therapies to acetaminophen for 14 weeks.

Exclusion Criteria:

* Subjects desiring escalation of analgesics for their current level of knee pain as determined by endorsement of the following statement: "Is your knee pain bad enough that you want to talk to your doctor about taking stronger pain medications?"
* Current use of opioids and/or Celebrex.
* Current use of an NSAID (not including ASA) for a painful condition in addition to knee OA.
* Contraindications to chronic NSAID use: current use of warfarin or antiplatelet agent other than ASA, allergy to any NSAID, active upper gastrointestinal ulceration in the previous 30 days, upper gastrointestinal bleeding in the past year, history of gastroduodenal perforation or obstruction, cardiovascular event within the past 6 months (myocardial infarction, cerebrovascular event, coronary-artery bypass graft, invasive coronary revascularisation, or new-onset angina), severe congestive heart failure (New York Heart Association class III-IV), evidence of serious anemia, hepatic, renal (including nephrotic syndrome), or blood coagulation disorders, and pregnancy.

***Though the investigators are proposing a RWT - and thus will not be initiating NSAID therapy - it would not be appropriate to continue NSAIDs (even when prescribed) in high-risk patients. The investigators acknowledge that these exclusion criteria limit generalizability, but the investigators feel justified to ensure subjects' safety.***

* Previous hyaluronic acid knee injections (within 6 months) or corticosteroid knee injections (within 3 months).
* Scheduled knee hyaluronic acid or corticosteroid injections, arthroscopy, or knee surgery.
* Co-morbid conditions that include the following: known other causes of arthritis (infectious arthritis, rheumatoid arthritis, connective tissue disease, or psoriatic arthritis), gout or pseudogout attack within the last 12 months, peripheral neuropathy or cardiopulmonary disease that limits walking more than knee pain, bone metastases or Paget's disease involving the lower extremities, and history of drug or alcohol abuse within the past 2 years, bilateral knee replacements or knee pain in the replaced knee only.
* Current involvement in litigation or receiving workmen's compensation.
* Hearing, cognitive impairment or mental illness, as determined by chart review that would preclude participation in a CBT program.
* For Women of Childbearing Age: Must not currently be pregnant, agree to avoid getting pregnant during the course of the study and should inform the study team if pregnancy occurs at any time during study participation.
* Previous meloxicam use discontinued due to lack of effective symptom relief
* Contraindications to prolonged NSAID use, per PI discretion.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490 (Actual)
Dates: Start 2013-09-02 (Actual); Primary Completion 2018-10-05 (Actual); Study Completion 2018-10-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - Providence VA Medical Center, Providence, RI, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goulet JL, Buta E, Brennan M, Heapy A, Fraenkel L. Discontinuing a non-steroidal anti-inflammatory drug (NSAID) in patients with knee osteoarthritis: Design and protocol of a placebo-controlled, noninferiority, randomized withdrawal trial. Contemp Clin Trials. 2018 Feb;65:1-7. doi: 10.1016/j.cct.2017.11.020. Epub 2017 Dec 2. PMID 29198731
- [Derived] Fraenkel L, Buta E, Suter L, Dubreuil M, Levy C, Najem C, Brennan M, Corn B, Kerns R, Goulet J. Nonsteroidal Anti-inflammatory Drugs vs Cognitive Behavioral Therapy for Arthritis Pain: A Randomized Withdrawal Trial. JAMA Intern Med. 2020 Sep 1;180(9):1194-1202. doi: 10.1001/jamainternmed.2020.2821. PMID 32702101

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 490 participants were enrolled and underwent the run-in; 364 (74%) participants remained eligible at the end of the run-in period and were randomized: 180 to placebo followed by CBT and 184 to meloxicam.
Groups:
- Placebo Followed by CBT: Eligible subjects will be randomized to Meloxicam 15 mg po QD vs placebo
  Cognitive Behavioral Therapy (CBT): Subjects originally assigned to placebo will receive cognitive behavioral therapy for 10 weeks
- Active Treatment With Meloxicam: Eligible subjects will be randomized to Meloxicam 15 mg po QD vs placebo
  Meloxicam 15 mg po QD: Eligible subjects will be take Meloxicam 15 mg po QD
Period: Overall Study
Arm/Group | Placebo Followed by CBT | Active Treatment With Meloxicam
Started | 180 | 184
Completed | 173 | 178
Not Completed | 7 | 6

BASELINE CHARACTERISTICS:
Population: 490 participants were enrolled and underwent the run-in; 364 (74%) participants remained eligible at the end of the run-in period and were randomized: 180 to placebo followed by CBT and 184 to meloxicam.
Groups:
- Placebo: Participants in Placebo (CBT) Arm
- Meloxicam: Participants in Meloxicam Arm
- Total: Total of all reporting groups
Arm/Group | Placebo | Meloxicam | Total
Number analyzed (Participants) | 180 | 184 | 364
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (11.8) | 58.5 (10.0) | 58.4 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 20 | 39
  Male | 161 | 164 | 325
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 120 | 112 | 232
  Non-Hispanic Black | 45 | 51 | 96
  Hispanic | 9 | 8 | 17
  Other | 6 | 13 | 19
WOMAC Pain [Mean (Standard Deviation); unit: units on a scale] — scores range from 0 to 20 with higher scores reflecting worse pain
  units on a scale | 5.4 (3.8) | 5.9 (3.9) | 5.6 (3.8)
WOMAC disability [Mean (Standard Deviation); unit: units on a scale] — scores range from 0 to 68, with higher scores indicating worse functional limitation
  units on a scale | 17.5 (12.1) | 17.9 (11.9) | 17.7 (12.0)

OUTCOME MEASURES:

1. Primary Outcome: Primary Endpoint: WOMAC Pain Score (Likert Scale Version) at 4 Weeks
Description: The WOMAC pain score has a possible score range of 0-20 for Pain and higher scores indicate worse pain. The WOMAC pain scale consists of 5 questions that ask about pain during walking, stair use, lying in bed at night, sitting, and standing. Each question is scored on a 5-point scale, where 0 = None, 1 = Mild pain, 2 = Moderate pain, 3 = Severe pain, and 4 = Very severe pain. Total pain scores range from 0 to 20 with higher scores reflecting worse pain. The WOMAC also includes a lower extremity disability scale. Both the pain scale and disability scale (17 items) can be analyzed separately.
Time Frame: 4 Weeks
Population: The WOMAC pain score was available for 84% (152/180) of participants in the placebo group and 92% (169/184) of participants in the meloxicam group four weeks post-randomization.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Placebo Followed by CBT: Participants in Placebo (CBT) Arm
Arm/Group | Placebo Followed by CBT | Meloxicam
Number analyzed (Participants) | 152 | 169
units on a scale | 8.08 (0.3) | 6.73 (0.28)

2. Secondary Outcome: Area Under the Curve (AUC) of the WOMAC Pain Scale Score Over 14 Weeks
Description: The AUC is a commonly used measure that combines multiple measurements over a specific time interval into a single index. The AUC provides a single score that quantifies each participant's total WOMAC score across the repeated measurements. The AUC is valid regardless of increases or decreases in reported pain over time. In this case, the possible range is 0-20, with higher scores indicating worse pain.
Time Frame: 14 Weeks
Population: Those with no post-randomization pain measurements (n= 5 in meloxicam group, n= 4 in placebo) were excluded from all analyses of pain, leaving 355 (98%) participants for this analysis.
Measure: Mean (Standard Error); unit: units on a scale*week
Arm/Group | Placebo | Meloxicam
Number analyzed (Participants) | 176 | 179
units on a scale*week | 7.48 (0.21) | 6.43 (0.21)

3. Secondary Outcome: Lower Extremity Disability
Description: Lower extremity disability: Lower extremity functional outcomes will be measured using the WOMAC disability scale. The physical disability scale contains 17 items that assess the amount of difficulty subjects say they have with climbing stairs, rising from a chair, walking, and other activities of daily living. Responses are measured and scored in the same way as the pain scale. The WOMAC lower extremity disability score has a possible score range of 0-68 and higher scores indicate worse functional limitation.
Time Frame: 14 weeks
Population: WOMAC lower extremity disability scores were available in 336 (92%) participants at the end of Phase 2.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Active Treatment: Eligible subjects will be randomized to Meloxicam 15 mg po QD vs placebo
  Meloxicam 15 mg po QD: Eligible subjects will be take Meloxicam 15 mg po QD
Arm/Group | Active Treatment | Placebo
Number analyzed (Participants) | 160 | 176
score on a scale | 18.8 (0.9) | 19.7 (0.9)

4. Secondary Outcome: Global Impression of Change
Description: A balanced 5-point scale (rated 1 = Much better to 5 = Much worse) asking subjects to rate their change (if any) in pain since starting the study. The possible range of scores is 1 to 5.
Time Frame: 14 weeks
Population: Global impression of change was available in 336 (92%) participants at the end of Phase 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Meloxicam
Number analyzed (Participants) | 160 | 176
score on a scale | 2.15 (0.08) | 2.30 (0.08)

5. Secondary Outcome: Adherence to Study Medication (Assessed in Weeks Adherent)
Description: * Over the past week, how many days did you use the study drug for your knee pain?
  * Over the past week, how many days did you use Tylenol or acetaminophen for your knee pain?
  * Over the past week, how many days did you use other medications that were prescribed by one of your doctors for your knee pain?
  * Over the past week, how many days did you use other medications, creams or supplements that you got without a prescription for your knee pain?
  * Over the past week, how many days did you use any medications for a different problem or type of pain (e.g. headache)? Results reported as percentage of study weeks with perfect participant adherence to study medications, with higher percentages indicating higher adherence.
Time Frame: Weekly, for duration of observation period (14 weeks)
Population: All eligible subjects with any adherence data reported.
Measure: Median (Inter-Quartile Range); unit: Weeks Adherent
Arm/Group | Placebo | Active Treatment
Number analyzed (Participants) | 180 | 184
Weeks Adherent | 4 [3 to 4] | 13 [11 to 14]

6. Secondary Outcome: Adherence to Study Medication (Assessed in % of Weeks With Perfect Adherence)
Description: as for outcome 5
Time Frame: Weekly, for duration of observation period (14 weeks)
Population: All eligible subjects with any adherence data reported.
Measure: Number; unit: % weeks with perfect adherences
Arm/Group | Active Treatment | Placebo
Number analyzed (Participants) | 184 | 180
% weeks with perfect adherences | 87 | 91

ADVERSE EVENTS:
Time Frame: Adverse event data were collected through study completion, an average of 14 weeks. After 2-week run-in period where all subjects replaced their current NSAID with the study drug (meloxicam 15mg per day), remaining eligible subjects participated in 4-week, double-blind, placebo-controlled, non-inferiority randomized withdrawal trial (RWT). After 4 weeks, subjects in the meloxicam arm continued study drug. Subjects in the placebo arm stopped the placebo and participated in a 10-week CBT program.
Description: All related adverse events were identified by study coordinator or study therapist during the time when subject participates in the study. Any serious adverse events and unanticipated problems involving risks to subjects and others were reported immediately to the study PI and within 24 hrs to the VA Central Institutional Review Board (IRB). The reporting processes, as listed in the VA Central IRB Table of Reporting Requirements, was followed.
Arm/Group | Placebo | Meloxicam
All-Cause Mortality (participants affected / at risk) | 0/180 | 0/184
Serious Adverse Events (participants affected / at risk) | 3/180 | 4/184
Other Adverse Events (participants affected / at risk) | 0/180 | 0/184
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=180) | Meloxicam (N=184)
Bleeding hemorrhoid (Gastrointestinal disorders) | 0 (0) | 1 (1) — Patient represented with bleeding hemorrhoid requiring surgery and discontinuation of study drug (Meloxicam).
Chest Pain (Cardiac disorders) | 1 (1) | 2 (2) — Chest pain; one patient occurrence resolved without work-up; one resulted in need for cardiac cath; one resulted in coronary artery bypass graft surgery (CABG) and withdrawal from study
ischemic stroke (Vascular disorders) | 1 (1) | 0 (0) — Pt suffered ischemic stroke. Had been randomized to and taking placebo and had not taken Meloxicam for the past month. Pt withdrawn from Study per his request.
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) — Patient presented to emergency department (ED) with shortness of breath (SOB)/chest pain in Afib but discharged in sinus rhythm and was placed on Coumadin for 7days; study medication held as long as coumadin therapy was continued.
Arm celluitis (Infections and infestations) | 0 (0) | 1 (1) — Patient with prior breast cancer and axially node resection presented with arm swelling/redness and treated for infectious cellulitis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-06-28): https://cdn.clinicaltrials.gov/large-docs/13/NCT01799213/Prot_SAP_000.pdf